CLINICAL TRIAL: NCT01850680
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety and Tolerability of Subcutaneously Administered Sarilumab in Japanese Patients With Rheumatoid Arthritis Receiving Concomitant Methotrexate
Brief Title: Single Ascending Dose Study of Safety and Tolerability of Sarilumab and Methotrexate in Japanese Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDU13402; U1111-1134-0048 (Other: UTN)
Record Dates: First submitted 2013-05-01; First posted 2013-05-09 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sarilumab (SAR153191, REGN88) Dose 1 (Experimental): First dose of Sarilumab in a single SC injection. Methotrexate (stable dose) and folic acid are continued as background therapy
  Interventions: Drug: sarilumab SAR153191 (REGN88); Drug: methotrexate; Drug: folic acid
- Sarilumab (SAR153191, REGN88) Dose 2 (Experimental): Second dose of Sarilumab in a single SC injection. Methotrexate (stable dose) and folic acid are continued as background therapy
  Interventions: Drug: sarilumab SAR153191 (REGN88); Drug: methotrexate; Drug: folic acid
- Sarilumab (SAR153191, REGN88) Dose 3 (Experimental): Third dose of Sarilumab in a single SC injection. Methotrexate (stable dose) and folic acid are continued as background therapy
  Interventions: Drug: sarilumab SAR153191 (REGN88); Drug: methotrexate; Drug: folic acid
- Sarilumab (SAR153191, REGN88) Dose 4 (Experimental): Fourth dose of Sarilumab in a single SC injection. Methotrexate (stable dose) and folic acid are continued as background therapy
  Interventions: Drug: sarilumab SAR153191 (REGN88); Drug: methotrexate; Drug: folic acid
- Placebo Dose 5 (Placebo Comparator): Placebo to match Sarilumab (SAR153191, REGN88) in a single SC injection. Methotrexate (stable dose) and folic acid are continued as background therapy
  Interventions: Drug: placebo; Drug: methotrexate; Drug: folic acid

INTERVENTIONS:
Drug: sarilumab SAR153191 (REGN88) — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Sarilumab (SAR153191, REGN88) Dose 1; Sarilumab (SAR153191, REGN88) Dose 2; Sarilumab (SAR153191, REGN88) Dose 3; Sarilumab (SAR153191, REGN88) Dose 4
Drug: placebo — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Placebo Dose 5
Drug: methotrexate — Pharmaceutical form:capsule Route of administration: oral
Drug: folic acid — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

To assess the safety and tolerability of a single dose of subcutaneously administered sarilumab in Japanese patients with rheumatoid arthritis (RA) who are receiving concomitant treatment with methotrexate.

Secondary Objective:

To assess the pharmacokinetic profile of a single subcutaneous (SC) dose of sarilumab in Japanese RA patients.

DETAILED DESCRIPTION:
Total study duration per patient is up to 88 days

1. Screening: 3 to 28 days
2. Treatment: 1 day
3. Follow-up: 57± 3 days after dosing

ELIGIBILITY:
Inclusion criteria:

1. Male or female Japanese who are 20 to 65 years of age
2. Diagnosis of rheumatoid arthritis (RA) ≥ 3 months duration
3. Treated for a minimum of 8 weeks with Methotrexate (MTX) and with a stable dose of MTX (6-16 mg/week) for a minimum of 4 weeks prior to the screening visit

Exclusion criteria:

1. Autoimmune or inflammatory systemic or localized joint disease other than RA
2. Women of a positive pregnancy test
3. Latent or active tuberculosis
4. Prior treatment with anti-interleukin-6 (anti-IL-6) or anti-interleukin-6 receptor (IL-6R) antagonist
5. Treatment with anti-TNF agents, as follows:

   1. Etanercept: within 28 days prior to randomization
   2. Infliximab, adalimumab, golimumab, certolizumab pegol: within 42 days prior to randomization
6. Received any live, attenuated vaccine within 3 months prior to the randomization visit (eg, varicella-zoster, oral polio, rubella vaccines)
7. Significant concomitant illness such as, but not limited to, cardiovascular, renal, neurological, endocrinological, gastrointestinal, hepato-biliary, metabolic, pulmonary or lymphatic disease that would adversely affect the patient's participation in the study.
8. Received surgery within 4 weeks prior to the screening visit or planned surgery during the study
9. History of a systemic hypersensitivity reaction

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Assessment of safety parameters (adverse events, laboratory data, vital signs, and ECG) | Up to 88 days or end-of-study (EoS)
Assessment of the occurrence of anti-sarilumab antibodies | Day 1, Day 15, Day 29, Day 57
Assessment of the titer of anti-sarilumab antibodies | Day 1, Day 15, Day 29, Day 57

SECONDARY OUTCOMES:
Assessment of PK parameter - maximum concentration (Cmax) | At each visit, up to 88 days
Assessment of PK parameter - area under curve (AUC) | At each visit, up to 88 days
Assessment of PK parameter - time to maximum concentration (tmax) | At each visit, up to 88 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Japan (2):
  - Investigational Site Number 392001, Sendai
  - Investigational Site Number 392002, Sendai